CLINICAL TRIAL: NCT06216769
Title: Comparison Between Continuous Oral Anticoagulation Versus Pill-in-the-POCKET Oral AntiCoagulation Strategy Guided by Continuous Rhythm Monitoring Using Implantable Loop Recorder After Atrial Fibrillation Catheter Ablation
Brief Title: Pill-in-the-POCKET Oral Anticoagulation Strategy After AF Catheter Ablation
Acronym: POCKET-OAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Samjin Pharmaceutical Co., Ltd. (Industry); Medtronic Korea Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Eue-Keun Choi, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2304-038-1420
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; direct oral anticoagulant; catheter ablation; implantable loop recorder; continuous cardiac rhythm monitor
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-interrupted group (Active Comparator): Anticoagulation is continued regardless of atrial fibrillation recurrence.
  Interventions: Drug: Rivaroxaban
- PIP anticoagulation group (Experimental): Anticoagulation continuation will be determined based on the rhythm monitored by ILR. If atrial fibrillation persists more than 6 hours a day, anticoagulation should be started at that point on and continued for four weeks. Anticoagulation can be prescribed even in case of less-than-6-hour cumulative atrial fibrillation burden if the investigator decides that the anticoagulation is necessary.
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Rivaroxaban — Those in the non-interrupted anticoagulation group, anticoagulation is continued regardless of atrial fibrillation recurrence.
  Those in the pill-in-the POCKET anticoagulation group will receive direct oral anticoagulation only if they have atrial fibrillation recur over 6 hours.

SUMMARY:
The clinical benefit of pill-in-the-POCKET anticoagulation after atrial fibrillation catheter ablation remains uncertain. We aimed to evaluate the clinical benefit and safety of pill-in-the-POCKET anticoagulation after atrial fibrillation catheter ablation by randomizing into two groups: non-interrupted anticoagulation after the procedure and anticoagulation based on atrial fibrillation recurrence confirmed by implantable loop recorders.

DETAILED DESCRIPTION:
Atrial fibrillation significantly increases the risk of thromboembolic complications, including stroke. Accordingly, current atrial fibrillation treatment guidelines recommend lifelong prescription of anticoagulants if the CHA2DS2-VASc score is 2 (for males) or 3 (for females) or higher (Class IA). With the recent advances in rhythm control treatment through catheter ablation in atrial fibrillation patients, increasing concerns are being raised about the need to continue anticoagulation after successful catheter ablation. However, current guidelines still require continued anticoagulation based on the baseline CHA2DS2-VASc score regardless of sinus conversion after atrial fibrillation catheter ablation.

A recently published observational study demonstrated that the risk of stroke was reduced by less than 0.7% per year in patients who discontinued anticoagulants after successful catheter ablation. Subsequent meta-analysis studies similarly suggested that anticoagulant discontinuation could be safe in patients whose rhythm was restored to sinus rhythm through catheter ablation. In addition, it was confirmed that anticoagulant discontinuation after catheter ablation was associated with only a 0.6% increase in the risk of thromboembolism as opposed to a 1.8% decrease in the risk of severe bleeding, such as intracranial hemorrhage and respiratory bleeding. Similar findings were also confirmed from large-scale non-randomized studies. However, there is still a lack of large-scale randomized study findings to support that anticoagulant discontinuation is appropriate in atrial fibrillation who are successful converted to sinus rhythm after catheter ablation.

Two single-arm pilot studies have been published about pill-in-the-pocket (PIP) anticoagulation. One is the REACT.COM (Rhythm Evaluation for Anticoagulation With Continuous Monitoring), and the other is the TACTIC-AF (Tailored Anticoagulation for Non-Continuous Atrial Fibrillation). In the above studies, continuous remote monitoring was performed using insertable cardiac monitors, dual-chamber pacemakers, or defibrillators. If atrial fibrillation persisted over a certain period during monitoring, anticoagulation was resumed for 30 days. This approach reduced the use of anticoagulants by 94% in the REACT.COM by resuming anticoagulation when atrial fibrillation recurrence persisted longer than 1 hour. TACTIC-AF observed a 75% reduction in time on anticoagulation using a threshold of 6 minutes or total burden >6 h/d.

Conventionally, recurrence of atrial fibrillation has been confirmed through 12-lead electrocardiogram (ECG) or adhesive 24-hour (or 3-day, 7-day, 2-week) ECG monitoring. However, these methods are limited by the inability to continuously assess the exact atrial fibrillation burden during the follow-up period. As an alternative to this, implantable loop recorders (ILR) enabled with continuous heart rhythm monitoring have recently been widely used in clinical practice. These implantable loop recorders have shown desirable performance in measuring atrial fibrillation recurrence and burden. However, few studies have evaluated the role of continuous rhythm monitoring in guiding OAC in patients with AF.

This study is aimed to evaluate clinical benefits, including the appropriateness, efficacy, and safety of pill-in-the-POCKET anticoagulation, and establish its cost-effectiveness by comparing the incidence of major clinical events after randomization of atrial fibrillation patients scheduled to undergo catheter ablation into two groups: non-interrupted anticoagulation after the procedure and resumed anticoagulation based on atrial fibrillation recurrence confirmed by implantable loop recorders.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are scheduled to undergo atrial fibrillation catheter ablation due to atrial fibrillation refractory to antiarrhythmic drug treatment.
2. Patients with non-gender CHA2DS2-VASc score 1-4.
3. Patients who are taking direct oral anticoagulants (rivaroxaban, dabigatran, apixaban, edoxaban) and further plan taking them life-long to prevent stroke caused by atrial fibrillation.
4. Patients aged 19-89 (inclusive) who voluntarily sign the informed consent form.

Exclusion Criteria:

1. Patients with a stroke/transient ischemic attack history.
2. Patients with underlying diseases and bleeding findings contraindicated to anticoagulation (e.g., coagulation disorders, bleeding conditions, significant gastrointestinal bleeding within 6 months of enrollment, history of intracranial/intraocular/nontraumatic bleeding, thrombolysis within 48 hours of study enrollment).
3. Patients who are contraindicated to anticoagulants other than those listed above.
4. Patients who are hemodynamically unstable at the time of study enrollment: cardiogenic shock, treatment-unresponsive ventricular arrhythmia, or congestive heart failure (NYHA class IV) at the time of randomization.
5. Patients with underlying severe anemia (hemoglobin <8 g/dL at baseline) or a transfusion history within four weeks before visit 1.
6. Patients with underlying severe thrombocytopenia (platelet count <50,000/mm3)
7. The patient is under dialysis or chronic renal failure (creatinine clearance <15ml/min)
8. The patient has severe liver disease (variceal bleeding, ascites, hepatic encephalopathy, or jaundice).
9. The patient has a contraindication to the implantation of an implantable loop recorder (ILR) (such as limited immunocompetence or a wound-healing disorder).
10. The patient has severe valvular disease (valvular prosthesis, mitral valve repair; rheumatic mitral stenosis is excluded irrespective of the severity of the disease).
11. The patient has a non-arrhythmic condition necessitating long-term oral anticoagulation.
12. Hypertrophic cardiomyopathy
13. The patient is deemed high risk for non-cardioembolic stroke (i.e. significant carotid artery disease).
14. Patients who are taking warfarin or coumadin.
15. Patients who are taking dual antiplatelet agents.
16. Patients with a history of Cox-Maze surgery or atrial fibrillation catheter ablation for atrial fibrillation treatment.
17. Pregnancy, breastfeeding, or women of childbearing age who refuse to use a highly effective and medically acceptable form of contraception throughout the study. *

    * Medically acceptable contraceptives include condoms, injectable or implantable contraceptives, intrauterine devices, and oral contraceptives.
18. Known or suspected malignancy with a history of chemotherapy within 1 year.
19. The patient has previously implanted cardiac implantable electronic devices or ILR.
20. Patients with a history of left atrial appendage occlusion or left atrial appendage closure.
21. The patient is participating in another randomized clinical trial and is under follow-up observation.

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite of ischemic stroke, transient ischemic attack, other systemic embolism, bleeding (major, clinically relevant), all-cause death | up to 24 months

SECONDARY OUTCOMES:
Composite of thromboembolic events (ischemic stroke, transient ischemic attack, systemic embolism) | up to 24 months
Composite of bleeding events events (major bleeding and clinically relevant non-major bleeding) | up to 24 months
Individual components of the primary endpoint. | up to 24 months
  Any ischemic stroke, any transient ischemic attack, any systemic embolism, any major bleeding, any clinically relevant non-major bleeding, any death
All bleeding (major, clinically relevant non-major bleeding, and minor bleeding) | up to 24 months
Recurrence of any atrial arrhythmia lasting longer than 2 minutes (atrial arrhythmia: atrial fibrillation/atrial tachycardia) | up to 24 months
Atrial arrhythmia burden (%) between 3 and 24 months after catheter ablation | up to 24 months
Quality of Life scores assessed by Atrial Fibrillation Effect on QualiTy-of-life(AFEQT) questionnaire at baseline (preoperative) and at the end of 24 months, respectively | up to 24 months
Cognitive function assessed by Korea-Montreal Cognitive Assessment (K-MoCA) score questionnaire at baseline (preoperative) and at the end of 24 months, respectively | up to 24 months
Change in treatment according to ILR results | up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Passman R, Leong-Sit P, Andrei AC, Huskin A, Tomson TT, Bernstein R, Ellis E, Waks JW, Zimetbaum P. Targeted Anticoagulation for Atrial Fibrillation Guided by Continuous Rhythm Assessment With an Insertable Cardiac Monitor: The Rhythm Evaluation for Anticoagulation With Continuous Monitoring (REACT.COM) Pilot Study. J Cardiovasc Electrophysiol. 2016 Mar;27(3):264-70. doi: 10.1111/jce.12864. Epub 2015 Nov 23. PMID 26511221
- [Background] Waks JW, Passman RS, Matos J, Reynolds M, Thosani A, Mela T, Pederson D, Glotzer TV, Zimetbaum P. Intermittent anticoagulation guided by continuous atrial fibrillation burden monitoring using dual-chamber pacemakers and implantable cardioverter-defibrillators: Results from the Tailored Anticoagulation for Non-Continuous Atrial Fibrillation (TACTIC-AF) pilot study. Heart Rhythm. 2018 Nov;15(11):1601-1607. doi: 10.1016/j.hrthm.2018.06.027. Epub 2018 Jul 6. PMID 29981863
- [Background] Hindricks G, Pokushalov E, Urban L, Taborsky M, Kuck KH, Lebedev D, Rieger G, Purerfellner H; XPECT Trial Investigators. Performance of a new leadless implantable cardiac monitor in detecting and quantifying atrial fibrillation: Results of the XPECT trial. Circ Arrhythm Electrophysiol. 2010 Apr;3(2):141-7. doi: 10.1161/CIRCEP.109.877852. Epub 2010 Feb 16. PMID 20160169
- [Background] Karasoy D, Gislason GH, Hansen J, Johannessen A, Kober L, Hvidtfeldt M, Ozcan C, Torp-Pedersen C, Hansen ML. Oral anticoagulation therapy after radiofrequency ablation of atrial fibrillation and the risk of thromboembolism and serious bleeding: long-term follow-up in nationwide cohort of Denmark. Eur Heart J. 2015 Feb 1;36(5):307-14a. doi: 10.1093/eurheartj/ehu421. Epub 2014 Nov 3. PMID 25368205
- [Background] Themistoclakis S, Corrado A, Marchlinski FE, Jais P, Zado E, Rossillo A, Di Biase L, Schweikert RA, Saliba WI, Horton R, Mohanty P, Patel D, Burkhardt DJ, Wazni OM, Bonso A, Callans DJ, Haissaguerre M, Raviele A, Natale A. The risk of thromboembolism and need for oral anticoagulation after successful atrial fibrillation ablation. J Am Coll Cardiol. 2010 Feb 23;55(8):735-43. doi: 10.1016/j.jacc.2009.11.039. PMID 20170810